CLINICAL TRIAL: NCT04918862
Title: A Comparative Study of 1mg and 3 mg of Granisetron in the Prevention of Postoperative Nausea and Vomiting in Strabismus Ophthalmic Surgeries During General Anesthesia
Brief Title: A COMPARATIVE STUDY BETWEEN 1MG AND 3 MG OF GRANISETRON IN THE PREVENTION OF POSTOPERATIVE NAUSEA AND VOMITING IN STRABISMUS OPHTHALMIC SURGERIES DURING GENERAL ANESTHESIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Mohamed Yousry Mohamed (Unknown); Tamer Fayez Safan (Unknown); Tamer Mohamed Khair (Unknown); Mohamed, Ahmed A., M.D. (Individual); Islam Mohamed Sayed (Unknown)
Responsible Party: Principal Investigator, Ahmed Abdalla, Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MS-380-2020
Record Dates: First submitted 2021-05-20; First posted 2021-06-09 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: 1mg Vs 3 mg of Granisetron
MeSH Terms: interventions — Granisetron

STUDY DESIGN:
Intervention Model Description: 210 patients were recruited and allocated randomly to receive either granisetron 1.0mg (n =105) or granisetron 3.0mg (n =105). The two groups were compared regarding: demographic data of the patients, hemodynamic parameters including mean arterial pressure and heart rate and percentage of patients with no complain of postoperative nausea and vomiting at first 24 hours.
Who Masked: Participant
Masking Description: Computer-generated sequence will be used for randomization and opaque envelopes will be used for concealment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Granisetron 1 mg (Active Comparator): Granisetron 1 mg: 105 patients received 1mg granisetron
  Interventions: Drug: Granisetron
- Granisetron 3 mg (Active Comparator): Granisetron 3 mg: 105 patients received 3mg granisetron
  Interventions: Drug: Granisetron

INTERVENTIONS:
Drug: Granisetron — 210 patients were enrolled, divided into two groups [Granisetron 1 mg: 105 patients received 1mg granisetron, Granisetron 3 mg: 105 patients received 3mg granisetron]. The two groups were compared in demographic characteristics (age, gender, weight, and height), hemodynamic parameters (MAP and HR), and duration of surgery
  Other Names: Granisetron in the prevention of postoperative nausea and vomiting in strabismus ophthalmic surgeries during general anesthesia.

SUMMARY:
Investigators aim to determine the optimal dose of granisetron in strabismus ophthalmic surgeries under general anesthesia to prevent postoperative nausea and vomiting

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) are common and distressing symptoms after surgery under general anesthesia. Despite advances in balanced anesthesia in recent decades, PONV can result in delayed discharge from the Post-Anesthesia Care Unit (PACU) recovery room, unexpected hospitalization and increase in medical costs.

The latest class of antiemetic for the prevention and treatment of PONV are the serotonin receptor antagonists (ondansetron, granisetron). These antiemetics do not have the negative effects of the older generations. Headache and dizziness are the main adverse effects of the serotonin receptor antagonists in the dosages used for PONV .

The FDA approved dose for the prevention of PONV is 1mg. This is based on a dose range study from Wilson and associates in which 0.1, 1.0, and 3.0 mg were associated with risk ratios for postoperative vomiting. The majority of studies on granisetron suggest that 3mg is superior to 1mg for the prevention of PONV, but those were published by a single center and there have been serious concerns about the validity of the data. In previous studies done on elective open abdominal surgery or vaginal hysterectomy but not in strabismus ophthalmic surgeries.

The ocular surgery associated with the highest incidence of PONV is strabismus surgery up to 85%. Vomiting after surgery is more likely 2-8hours than immediate postoperatively. Strabismus is a day case procedure and thus participants have to cope with emesis in the recovery room, or when traveling, or at home.

In this study, investigators compared two doses of granisetron in strabismus ophthalmic surgeries under general anesthesia

ELIGIBILITY:
Inclusion Criteria:

* • Adult patients > 18 years old.

  * ASA I and II.
  * Patients scheduled for strabismus surgery.

Exclusion Criteria:

* • ASA class > II.

  * Patients with known hypersensitivity or contraindication to any of the study medications.
  * Patients who had chronic nausea and vomiting or experienced retching, vomiting, moderate to severe nausea in the preoperative day.
  * Patients who had received an antiemetic drug in the preoperative day.
  * Patients with a body mass index ≥36.
  * Pregnant or breast feeding female patient.
  * Patients with gastrointestinal diseases.
  * Patients with a history of motion sickness, diabetes mellitus, and GIT pathology (gastritis, hematemesis, peptic ulcer).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-05-09 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
The percent of patients with total control of nausea and vomiting over the first 24 hrs postoperative | Up to 24 hours
  The percent of patients with total control of nausea and vomiting over the first 24 hrs postoperative

SECONDARY OUTCOMES:
Detection of the optimal dose of granisetrone | Up to 24 hours
  Detection of the optimal dose of granisetrone/mg
Detection of either attacks of nausea and vomiting occurred post operatively or not. • | Post operatively over the first 24 hrs postoperative .
  Detection of either attacks of nausea and vomiting occurred post operatively or not
Blood Pressure | Up to 24 hours
  Blood Pressure measurment mmHg
Heart Rate | Up to 24 hours
  Heart Rate measurment beat /minute

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Mohamed, M.D, Principal Investigator — Cairo University
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Till Submission